CLINICAL TRIAL: NCT04647669
Title: WHO Public Health Emergency "Solidarity" Clinical Trial for COVID-19 Treatments
Brief Title: World Health Organization (WHO) COVID-19 Solidarity Trial for COVID-19 Treatments
Acronym: SOLIDARITY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRD/ETH/20
Record Dates: First submitted 2020-10-15; First posted 2020-12-01 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; acalabrutinib; Interferon beta-1a; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Local Standard of Care (Placebo Comparator): Local Standard of Care
  Interventions: Other: Standard of Care
- Remdesivir (Active Comparator): Remdesivir (daily infusion for 10 days)
  Interventions: Drug: Remdesivir
- Acalabrutinib (Active Comparator): Acalabrutinib (orally twice daily for 10 days)
  Interventions: Drug: Acalabrutinib
- Interferon (Active Comparator): Interferon β1a(daily injection for 6 days).
  Interventions: Drug: Interferon beta-1a

INTERVENTIONS:
Drug: Remdesivir — 200 mg intravenous loading dose on Day 1, and 100mg intravenous once-daily for subsequent doses from Day 2 up to Day 10.
  Arms: Remdesivir
Drug: Acalabrutinib — 100 mg capsules twice daily every 12 h for 10 days taken with or without food.
  Arms: Acalabrutinib
Drug: Interferon beta-1a — Interferon ß-1a will be administered intravenously at the dose of 10 μg once daily for 6 days if oxygen dependent or subcutaneously at 44 ug Day 1, Day 3, and Day 6
  Arms: Interferon
Other: Standard of Care — Treatment according to local hospital protocol
  Arms: Local Standard of Care

SUMMARY:
In early 2020 there were no approved anti-viral treatments for COVID19 Infection. The SOLIDARITY trial is a multicentre adaptive international randomised trial sponsored by Word Health Organization to determine the efficacy of Remdesivir (daily infusion for 10 days), or Acalabrutinib (orally twice daily for 10 days), or Interferon β1a(daily injection for 6 days) compared with local standard of care in patients admitted to hospital for COVID19 infection on all-cause mortality, stratified by severity of disease at the time of randomisation. The major secondary outcomes are duration of hospital stay and time to first receiving ventilation (or intensive care).

DETAILED DESCRIPTION:
Terminology: The novel coronavirus-induced disease first described in 2019 in China is designated COVID-19 (or COVID), and the pathogen itself (an RNA virus) is SARS-coronavirus-2 (SARS-CoV-2).

Background: In early 2020 there were no approved anti-viral treatments for COVID, and WHO expert groups advised that four re-purposed drugs, Remdesivir, Lopinavir (given with Ritonavir, to slow hepatic degradation), Interferon (β1a), and hydroxychloroquine (HCQ) should be evaluated in an international randomised trial. In addition, WHO provided guidelines that local physicians may consider when COVID-19 is suspected on clinical management of severe acute respiratory infection. However, following an interim analyses, the interim results of HCQ vs standard of care and lopinavir/ritonavir vs standard of care from the Solidarity/Discovery trials, the Solidarity trial Executive Group decided to stop the HCQ and the Lopinavir/ritonavir arms on the 3rd of July, 2020 due to futility; leaving 3 arms, i.e., remdesivir, Interferon (β1a), and standard of care.

On the 6th of August 2020, due to a review of the rationale and clinical evidence, the Executive Group of the Steering Committee of the Solidarity trial recommended that a new arm should be opened in the Solidarity trial, to evaluate the clinical efficacy of Acalabrutinib.

Simplicity of procedures: To facilitate collaboration even in hospitals that have become overloaded, patient enrolment and randomisation (via the internet) and all other trial procedures are greatly simplified, and no paperwork at all is required. Once a hospital has obtained approval, electronic entry of patients who have given informed consent takes only a few minutes. At the end of it, the randomly allocated treatment is displayed on the screen and confirmed by electronic messaging.

Randomisation: Adults (age ≥18 years) recently hospitalised, or already in hospital, with definite COVID and, in the view of the responsible doctor, no contra-indication to any of the study drugs will be randomly allocated between

* Local standard of care alone, OR local standard of care plus one of
* Remdesivir (daily infusion for 10 days)
* Acalabrutinib (orally twice daily for 10 days)
* Interferon β1a(daily injection for 6 days).

Data reported before randomisation: Information is entered electronically on

* Country, hospital (from a list of approved hospitals) and randomising doctor
* Confirmation that informed consent has been obtained
* Patient identifiers, age and sex
* Patient characteristics (yes/no): current smoking, diabetes, heart disease, chronic lung disease, chronic liver disease, asthma, HIV infection, active tuberculosis.
* COVID-19 severity at entry (yes/no): shortness of breath, being given oxygen, already on a ventilator, and, if lungs imaged, major bilateral abnormality (infiltrations/patchy shadowing)
* Whether any of the study drugs are currently NOT AVAILABLE at the hospital.

Exclusion from study entry: Patients will not be randomised if, in the view of the randomising doctor, ANY of the AVAILABLE study drugs are contra-indicated (e.g., because of patient characteristics, chronic liver or heart disease, or some concurrent medication).

Changing management of study patients: At all times the patient's medical team remains solely responsible for decisions about that patient's care and safety. Hence, if the team decide that deviation from the randomly allocated treatment arm is definitely necessary, this should be done.

Follow-up: When patients die or are discharged, follow-up ceases and it is reported:

* Which study drugs were given (and for how many days)
* Whether ventilation or intensive care was received (and, if so, when it began)
* Date of discharge, or date and cause of death while still in hospital. If no report is received within 6 weeks of study entry, an electronic reminder is sent.

Drug safety: Suspected unexpected serious adverse reactions that are life-threatening (e.g., Stevens-Johnson syndrome, anaphylaxis, aplastic anaemia, or anything comparably uncommon and serious) must be reported within 24 hours of being diagnosed, without waiting for death or discharge.

Major outcomes: The primary outcome is all-cause mortality, subdivided by severity of disease at the time of randomisation. The major secondary outcomes are duration of hospital stay and time to first receiving ventilation (or intensive care).

Data monitoring: A global Data and Safety Monitoring Committee will keep the accumulating drug safety results and major outcome results under regular review.

Numbers entered: The larger the number entered the more accurate the results will be, but numbers entered will depend on how the epidemic develops. If substantial numbers get hospitalised in the participating centres, it may be possible to enter several thousand hospitalised patients with relatively mild disease and a few thousand with severe disease, but realistic, appropriate sample sizes could not be estimated at the start of the trial and will depend on the evolution of the epidemic.

Heterogeneity between populations: If a study treatment does affect outcome, then this effect could well differ between patients who had severe disease when randomised and those who had less severe disease. It could also differ between younger and older patients, or between patients in one or another country. If sufficient numbers are randomised, it may be possible to obtain statistically reliable treatment comparisons within each of several different countries or types of patient.

Adaptive design: The WHO may decide to add novel treatment arms while the trial is in progress. Conversely, the WHO may decide to discontinue some treatment arms, especially if the Global Data and Safety Monitoring Committee reports, based on interim analyses, that one of the trial treatments definitely affects mortality.

ELIGIBILITY:
Inclusion Criteria:

* consenting adults (age ≥18) hospitalised with definite COVID-19
* Patients without known allergy or contra-indications to any of the of the therapies and without anticipated transfer within 72 hours to a non- study hospital.
* Patients admitted to a collaborating hospital Exclusion Criteria
* AVAILABLE study drugs are contra-indicated (e.g., because of patient characteristics, chronic liver or heart disease, or some concurrent medication).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause Mortality | Number of days from hospital admission up to 28 days post discharge

SECONDARY OUTCOMES:
Duration of hospital stay | Number of days from hospital admission to discharge up to 28 days post admission
Time to first receiving ventilation | Number of days from hospital admission to day of receiving ventilatory support up to 28 days post admission
Time to admission to the intensive care unit | Number of days from hospital admission to day of admission to intensive care unit up to 28 days post admission

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Reid, Principal Investigator — University of the West Indies
Locations (1):
- Univeristy of the West Indies, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582